CLINICAL TRIAL: NCT01865604
Title: Impact of tDCS on Cerebral Autoregulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Agnes Flöel, Prof. Dr. med. Agnes Floeel, Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: tDCS_cVMR
Record Dates: First submitted 2012-12-18; First posted 2013-05-31 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Cerebral Microangiopathy; CADASIL; Migraine With Aura; ICA Stenosis
MeSH Terms: conditions — Cerebral Small Vessel Diseases; CADASIL; Migraine with Aura | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Anodal tDCS (Experimental): anaodal transcranial direct current stimulation
  Interventions: Device: Anodal tDCS
- Cathodal tDCS (Active Comparator): cathodal transcranial direct current stimulation
  Interventions: Device: Cathodal tDCS
- Sham tDCS (Sham Comparator): no stimulation
  Interventions: Device: sham tDCS

INTERVENTIONS:
Device: Anodal tDCS
  Arms: Anodal tDCS
Device: Cathodal tDCS
  Arms: Cathodal tDCS
Device: sham tDCS
  Arms: Sham tDCS

SUMMARY:
The aim of the study is to investigate whether there is a polarity-specific influence of tDCS on cerebral vasomotor reactivity monitored by transcranial doppler sonography.

ELIGIBILITY:
Inclusion Criteria:

1. severe cerebral Microangiopathy
2. NOTCH3 carrier
3. Migraine with aura (IHS Classification ICHD-II)
4. Stenosis >80%, ECST-Criteria

Exclusion Criteria:

* seizure disorder
* history of severe alcohol or drug abuse, psychiatric illness like severe depression, poor motivational capacity
* dementia

(1+2) history of stroke in past 3 months (3) migraine prophylaxis (4) contralateral stenosis >50%,

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-04; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Cerebral vasomotor reactivity assessed by transcranial Dopplersonography | on 3 days within 12 weeks
  comparing cerebral vasomotor reactivity at baseline and after anodal/cathodal/sham stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Flöel, Prof. MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Department of Neurology, Charité Universitätsmedizin Berlin, Berlin, State of Berlin, Germany